CLINICAL TRIAL: NCT01567891
Title: A Phase I/IIa, Open Label Clinical Trial Evaluating the Safety and Efficacy of Autologous T Cells Expressing Enhanced TCRs Specific for NY-ESO-1 in Patients With Recurrent or Treatment Refractory Ovarian Cancer.
Brief Title: CT Antigen TCR-redirected T Cells for Ovarian Cancer.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0011-001; 230612 (Other: Adaptimmune)
Record Dates: First submitted 2012-03-16; First posted 2012-03-30 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2018-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Cell Therapy; T Cell Therapy; NY-ESO-1; Immuno-oncology; Metastatic; Previously treated; T Cell Receptor
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): This is an open label clinical trial. Patients with the HLA-A201, HLA-A205, and/or HLA-A206 allele and whose tumor expresses the NY-ESO-1 tumor antigen will be eligible to receive NYESO-1c259 T cells.
  Interventions: Biological: NYESO-1c259 T cells

INTERVENTIONS:
Biological: NYESO-1c259 T cells — Cytoreductive chemotherapy followed by infusion with NYESO-1(C259) transduced autologous T cells. Patients will receive at least 1x10⁹ transduced cells, however the target dose for this protocol is for patients to receive 5x10⁹ transduced cells with a maximum possible dose of 6x10⁹ administered as a single intravenous (IV) infusion.

SUMMARY:
This study, will take a subject's "T cells" and "teach" them to be able to recognize and attack the ovarian cancer cells. This is done by putting in a gene or genetic material that will change how a subject's T cells work and hopefully get them to attack and kill ovarian cancer cells. These new T cells are called "engineered T cells" because the new gene is causing them to become directed toward the ovarian cancer cells rather than their usual targets. These are also called "gene-modified T cells". For subjects who have the HLA A2 tissue-type marker, the T cells would be engineered to recognize a substance called "NY-ESO-1". After putting this new gene in T cells (a procedure called "gene therapy") the investigators will grow the cells in the laboratory and give these cells back to subjects.

DETAILED DESCRIPTION:
This is an open label clinical trial. Patients with the HLA-A201, HLA-A205, and/or HLA-A206 allele and whose tumor expresses the NY-ESO-1 tumor antigen will be eligible to receive NY-ESO-1ᶜ²⁵⁹T. The trial is conducted entirely with outpatient procedures; however, patients may be hospitalized for the cytoreductive chemotherapy at the discretion of the investigator. Upon enrollment, patients will undergo leukapheresis for T cell collection, and their cells will be genetically engineered and expanded ex vivo. Seven days prior to receiving T-cells patients will undergo a cyclophosphamide conditioning regimen to potentiate the immunotherapy. The cell product will be infused as a single infusion (Day 0, typically Monday) to mitigate risks associated with unanticipated infusion reactions. Patients will be followed daily for the first week, weekly until 4 weeks, 8 weeks, and 12 weeks and then at 6 months and every 3 months until disease progression. Patients will undergo disease monitoring by MRI/CT scan (as appropriate for disease) at baseline, day 28, 8 weeks and 12 weeks, and months 6, and every 3 months until progression. Tumor biopsies will be taken at baseline, Week 8, and upon progression. In patients who have progressive disease following initial infusion but whose tumors continue to express NY-ESO-1, these patients may be eligible for a second infusion with redirected T cells. At disease progression, the interventional portion of the protocol ends and long term follow-up (LTFU) begins, in accordance with FDA regulations. LTFU occurs semiannually for up to 5 years post infusion and then annually thereafter for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of recurrent epithelial ovarian, primary peritoneal or fallopian tube carcinoma with refractory or platinum resistant disease and/or have received ≥ 2 lines of chemotherapy
* Age ≥ 18 years of age
* No significant immunodeficiency
* Have been informed of other treatment options
* Must be HLA A*0201, HLA-A*0205, and/or HLA-A*0206 positive by high resolution testing.
* Patient's tumor must be positive by histological assay for NY-ESO-1ᶜ²⁵⁹T, according to the screening algorithm as described in Section 3.3.1. Positive expression is defined as ≥ 50% of cells that are 2+ and/or 3+ by immunohistochemistry
* ECOG performance status of 0 or 1
* Life expectancy of > 4 months
* Prior therapies:

  1. prior immunotherapy, or prior investigational agents should be washed out 4 weeks before apheresis and must be completed 4 weeks prior to pre-infusion lymphodepletive chemotherapy.
  2. monoclonal antibody therapy must be completed at least 6 weeks prior to pre-infusion lymphodepletive chemotherapy
  3. All previous cytotoxic chemotherapy, monoclonal antibody therapy, immune therapy should be washed out 3 weeks before apheresis and must be completed at least 3 weeks prior to pre-infusion lymphodepletive chemotherapy.
  4. Systemic corticosteroid or other immunosuppressive therapy should be washed out 2 weeks before apheresis and must be completed at least 2 weeks prior to pre-infusion lymphodepletive chemotherapy
  5. Biologic or other approved molecular targeted small molecule inhibitors should be washed out 1 week before apheresis and must be completed at least 1 week prior to pre-infusion lymphodepletive chemotherapy.
  6. Any grade 3 or 4 -hematologic toxicity of previous therapy must have resolved to grade 2 or less prior to apheresis and any grade 3 or 4 toxicity must have resolved to grade 2 or less prior to pre-infusion lymphodepletive chemotherapy.
* Must have measurable disease as defined by RECIST 1.1.
* Must have adequate venous access for apheresis.
* Women of childbearing potential are requested to use acceptable methods of birth control for the duration of the study and until persistence of the study drug is no longer detected in the patient. This may be a period of several years. Methods for acceptable birth control include: condoms, diaphragm or cervical cap with spermicide, intrauterine device, and hormonal contraception. It is recommended that a combination of two methods be used.

Patients must have normal organ and marrow function as defined below:

* Leukocytes ≥ 3,000/mcL
* Absolute Neutrophil Count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin ≤ 1.5 ULN
* AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
* creatinine ≤ 2.0 mg/dL OR
* creatinine clearance > 60 mL/min for patients with creatinine levels above institutional normal
* Patient must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Currently receiving any other investigational agents
* Patients with active brain metastases. Patients with prior history of brain metastasis who have undergone local therapy (i.e. metastatectomy and/or radiation) and show no evidence of local recurrence or progression over the past 6 months are eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide or other agents used in the study
* Prior malignancy (except non-melanoma skin cancer) within 18 months of study entry NOTE: Patients must be in complete remission from prior malignancy in order to be eligible to enter the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g. interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to study entry. NOTE: Recent or current use of inhaled steroids is not exclusionary. If subjects are prescribed a brief course of oral corticosteroids, the use should be limited to less than 7 days. Use of steroids before apheresis and immune assessment blood draws should be discouraged as it will affect white blood cell function.
* Active infection with HIV, HBV or HCV
* Receipt of an experimental vaccine within 2 months or in the opinion of the Investigator is responding to an experimental vaccine given within 6 months, or has received any previous gene therapy using an integrating vector
* History of severe autoimmune disease requiring steroids or other immunosuppressive treatments
* Lack of availability of a patient for immunological and clinical follow-up assessment
* Evidence or history of significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, MD, PhD, Study Chair — Roswell Park Cancer Institute
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Institute, Stanford, California
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- NY-ESO-1ᶜ²⁵⁹T Cells Administered Intravenously: Participants who received cytoreductive chemotherapy followed by Lentivirus-mediated genetically engineered NY-ESO-1ᶜ²⁵⁹T (Target dose: 5 billion cells)
Period: Overall Study
Arm/Group | NY-ESO-1ᶜ²⁵⁹T Cells Administered Intravenously
Started | 9
Received T-cell | 6
Completed | 6
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Participants who received cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T
Groups:
- NY-ESO-1ᶜ²⁵⁹T: Participants who received cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T.
Arm/Group | NY-ESO-1ᶜ²⁵⁹T
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 58 [52 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Related to Study Treatment
Description: Number of Participants with Adverse Events related to study treatment
Time Frame: Up to 12 months
Population: Participants who received cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1ᶜ²⁵⁹T
Number analyzed (Participants) | 6
Participants | 5

2. Secondary Outcome: Tumor Response
Description: Number of participants with response as assessed by Immune-related Response Criteria (irRC)
Time Frame: Change from baseline, every 4 weeks until month 3 and then every 3 month until disease progression
Population: Participants who received cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1ᶜ²⁵⁹T
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Peak Persistence of Modified T-cells in the Peripheral Blood
Description: Measurement of NY-ESO-1ᶜ²⁵⁹T cells in blood
Time Frame: Days: 1, 2-4, weeks 1 to 4, Week 8, 12 and Month 6, then every 3 months thereafter until progression then during LTFU
Population: Participants who received NY-ESO-1ᶜ²⁵⁹T
Measure: Mean (Full Range); unit: copies of WPRE/mcg of genomic PBMC DNA
Groups:
- NY-ESO-1ᶜ²⁵⁹T: Participants who received NY-ESO-1ᶜ²⁵⁹T
Arm/Group | NY-ESO-1ᶜ²⁵⁹T
Number analyzed (Participants) | 6
copies of WPRE/mcg of genomic PBMC DNA | 85862.6 [27,310 to 169,753]

4. Secondary Outcome: Determine Functional Properties and Phenotype of Modified T-cells From Peripheral Blood.
Description: Percentage of CD4+pentamer+ or CD8+pentamer+ cells expressing LAG-3, PD-1, TIM-3 in the functionality of NY-ESO-1ᶜ²⁵⁹T cells in the manufactured product and post-treatment blood.
Time Frame: Weeks 4 and 8 post T-cell infusion
Measure: Number; unit: percentage of T cell sub population
Units Other Than Participants: T-cell sub population
Groups:
- Manufactured Product -Mean % CD4+Pentamer+; Week 4 Post-treatment- Mean % CD4+Pentamer+; Week 8 Post-treatment - Mean % CD4+Pentamer+; Manufactured Product - Mean % CD8+Pentamer+; Week 4 Post-treatment - Mean % CD8+Pentamer+; Week 8 Post-treatment - Mean % CD8+Pentamer+: Participants who received NY-ESO-1ᶜ²⁵⁹T
Arm/Group | Manufactured Product -Mean % CD4+Pentamer+ | Week 4 Post-treatment- Mean % CD4+Pentamer+ | Week 8 Post-treatment - Mean % CD4+Pentamer+ | Manufactured Product - Mean % CD8+Pentamer+ | Week 4 Post-treatment - Mean % CD8+Pentamer+ | Week 8 Post-treatment - Mean % CD8+Pentamer+
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Number analyzed (T-cell sub population) | 3 | 3 | 3 | 3 | 3 | 3
percentage of T cell sub population
  %LAG-3 | 4 | 3 | 0 | 3 | 0 | 0
  %PD-1 | 6 | 0 | 3 | 1 | 1 | 4
  %TIM-3 | 97 | 17 | 11 | 97 | 24 | 7

5. Secondary Outcome: Correlate NY-ESO-1 Expression in Tumor Tissue Before Treatment With Archival Tumor Tissue to Assess Impact of Therapy on Expression of NY-ESO-1 Protein
Description: NY-ESO-1 expression as determined by Histoscore (H score). Histoscore (0-300) represents the amount of NY-ESO-1 protein present in the tissue sample.
  H-Score formula:
  [1 × (% cells 1+) + 2 × (% cells 2+) + 3 × (% cells 3+)]
  (It is not clearly established if NY-ESO-1 H score has an association with prognosis.)
Time Frame: Screening and at Baseline
Population: Data is presented for 2 subjects, 4 subjects declined Baseline biopsy or biopsy wasn't collected due to safety concerns
Measure: Number; unit: H score
Groups:
- Subject 1; Subject 2: Participants who received NY-ESO-1ᶜ²⁵⁹T
Arm/Group | Subject 1 | Subject 2
Number analyzed (Participants) | 1 | 1
H score
  Screening/Archival | 50 | 100
  Baseline | 15 | 0

ADVERSE EVENTS:
Time Frame: Start of lymphodepletion to end of intervention phase (up to 12 months post T-cell infusion)
Description: Participants who received NY-ESO-1ᶜ²⁵⁹T
Arm/Group | NY-ESO-1ᶜ²⁵⁹T
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NY-ESO-1ᶜ²⁵⁹T (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (6)
Cytokine Release Syndrome (Immune system disorders) | 2 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (6)
Disease Progression (General disorders) | 1 (6)
Pancytopenia (Blood and lymphatic system disorders) | 1 (6)
Presyncope (Nervous system disorders) | 1 (6)
Pyrexia (General disorders) | 1 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NY-ESO-1ᶜ²⁵⁹T (N=6)
White blood cell count decreased (Investigations) | 6 (6)
Neutrophil count decreased (Investigations) | 5 (6)
Nausea (Gastrointestinal disorders) | 4 (6)
Abdominal Pain (Gastrointestinal disorders) | 3 (6)
Decreased appetite (Metabolism and nutrition disorders) | 3 (6)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (6)
Fatigue (General disorders) | 3 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (6)
Anemia (Blood and lymphatic system disorders) | 2 (6)
Ascites (Gastrointestinal disorders) | 2 (6)
Confusional state (Psychiatric disorders) | 2 (6)
Constipation (Gastrointestinal disorders) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 2 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Headache (Nervous system disorders) | 2 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Pyrexia (General disorders) | 2 (6)
Rash (Skin and subcutaneous tissue disorders) | 2 (6)
Sinus Tachycardia (Cardiac disorders) | 2 (6)
Alanine aminotransferase increased (Investigations) | 1 (6)
Anal incontinence (Gastrointestinal disorders) | 1 (6)
Anxiety (Psychiatric disorders) | 1 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (6)
Asparate aminotransferase increased (Investigations) | 1 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (6)
Blood alkaline phosphatase increased (Investigations) | 1 (6)
Blood creatinine increased (Investigations) | 1 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (6)
Chills (General disorders) | 1 (6)
Conjunctivitis (Immune system disorders) | 1 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (6)
Dizziness (Nervous system disorders) | 1 (6)
Facial Pain (General disorders) | 1 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (6)
Hypernatremia (Metabolism and nutrition disorders) | 1 (6)
Hypersensitivity (Immune system disorders) | 1 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (6)
Hypotension (Vascular disorders) | 1 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (6)
Lymphademopathy (Blood and lymphatic system disorders) | 1 (6)
Lymphopenia (Blood and lymphatic system disorders) | 1 (6)
Malaise (General disorders) | 1 (6)
Mucosal infection (Infections and infestations) | 1 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (6)
Edema (General disorders) | 1 (6)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Presyncope (Nervous system disorders) | 1 (6)
Proteinuria (Renal and urinary disorders) | 1 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (6)
Renal failure (Renal and urinary disorders) | 1 (6)
Serum ferritin increased (Investigations) | 1 (6)
Stomatitis (Gastrointestinal disorders) | 1 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (6)
Troponin increased (Investigations) | 1 (6)
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Urinary tract infection (Infections and infestations) | 1 (6)
Vomiting (Gastrointestinal disorders) | 1 (6)
Vulvovaginal candidiasis (Infections and infestations) | 1 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT01567891/SAP_000.pdf
  • Study Protocol (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT01567891/Prot_001.pdf